CLINICAL TRIAL: NCT06465784
Title: Comparison Between Retrograde and Antegrade Ureteroscopic Laser Lithotripsy for Management of Medium Sized Proximal Ureteral Stones: A Randomized Prospective Study
Brief Title: Laser Lithotripsy for Ureteral Stones
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahmoud Helmy El saeed Hussein (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Helmy El saeed Hussein, Professor, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Urosurg./Ms/2023/0001
Record Dates: First submitted 2024-05-29; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Ureteric Stone
Keywords: laser treatment; ureteric stones; ureteroscope; retrograde; antegrade
MeSH Terms: conditions — Ureterolithiasis

STUDY DESIGN:
Intervention Model Description: laster lithotripsy for clearance of uretric stones
Who Masked: Participant, Outcomes Assessor
Masking Description: Used closed envelope method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrograde Ureteroscopic Laser Lithotripsy (Active Comparator): In this arm we used the retrograde ureteroscopic Laser lithotripsy to clear the uretric stones. After the end of the procedure, all patients were followed for stone free rate as the primary outcome
  Interventions: Procedure: Retrograde and Antegrade Ureteroscopic Laser Lithotripsy
- Antegrade Ureteroscopic Laser Lithotripsy (Active Comparator): In this arm we used the antegrade ureteroscopic Laser lithotripsy to clear the uretric stones. After the end of the procedure, all patients were followed for stone free rate as the primary outcome.
  Interventions: Procedure: Retrograde and Antegrade Ureteroscopic Laser Lithotripsy

INTERVENTIONS:
Procedure: Retrograde and Antegrade Ureteroscopic Laser Lithotripsy — Comparison Between Retrograde and Antegrade Ureteroscopic Laser Lithotripsy for Management of Medium Sized Proximal Ureteral Stones: A Randomized Prospective Study

SUMMARY:
Objectives: To present the outcomes of retrograde and antegrade ureteroscopic laser lithotripsy in the treatment of proximal ureteral stones ranging in size from 10 to 20 millimeters in diameter.

Patients and methods: From March 2023 to December 2023, 70 patients were included in this prospective randomized double-arm interventional study. Patients were divided into two groups: Group 1: (35 patients) had semi-rigid retrograde ureteroscopic laser lithotripsy and group 2: (35 patients) had semi-rigid antegrade ureteroscopic laser lithotripsy.

DETAILED DESCRIPTION:
The present study was conducted in Al-Azhar University Hospital (Damietta branch), urology department,at the period from March 2023 to December 2023. Seventy patients with symptomatic proximal medium sized ureteric stones were classified in two groups Retrograde Uretroscopic Laser Lithotripsy (group 1) and Antegrade Ureteroscopic Laser Lithotripsy (group 2) .

The preoperative-(patient- and stone-related), intraoperative- and postoperative- related parameters that might influence the perioperative course and short-term clinical outcomes were evaluated.

ELIGIBILITY:
Inclusion Criteria:

- Patients with medium-sized proximal ureteral stones (10-20 mm) situated between the ureteropelvic junction and the top edge of the L5 vertebral body; age 18-65 years

Exclusion Criteria:

* Pregnancy, bleeding disorders, morbid obesity (BMI > 35), patients with stenosis of the ureter, history of previous surgery on the ipsilateral ureter, patients with a simultaneous kidney stone requiring surgery, and patients with an active urinary tract infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Stone free rate | Direct after intervention
  number of patients reported complete clearance of stones after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Damietta Faculty of Medicine, Al-Azhar University, Damietta, Egypt., Damietta, Egypt

IPD SHARING:
Plan to Share IPD: No